CLINICAL TRIAL: NCT05367271
Title: The Efficacy of Botulinum Toxin to the Flexor Digitorum Brevis Versus Corticosteroid to the Plantar Fascia for the Treatment of Refractory Plantar Fasciitis: A Randomized-Controlled Trial
Brief Title: The Efficacy of Botulinum Toxin vs. Corticosteroid for the Treatment of Refractory Plantar Fasciitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Western Institute for Veterans Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00146615
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Plantar Fasciitis
Keywords: OnabotulinumtoxinA; Botulinum Toxin A; Plantar fasciitis; Corticosteroid
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Botulinum Toxins, Type A; Dexamethasone; Cortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin A (BTX-A) (Experimental): 20 units of Onabotulinum A in 200 µL of saline
  Interventions: Drug: Botulinum Toxin A
- Corticosteroid (Active Comparator): 1 mL of 4 mg/mL dexamethasone with 2 mL of 1% lidocaine OR 1 mL of 4 mg/mL dexamethasone, 1 mL of 2% lidocaine and 1 mL saline
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Botulinum Toxin A — 20 units of Onabotulinum A in 200 µL of saline injected into the flexor digitorum brevis via ultrasound-guidance
  Other Names: OnabotulinumtoxinA; BTX-A
  Arms: Botulinum Toxin A (BTX-A)
Drug: Dexamethasone — 1 mL of 4 mg/mL dexamethasone with 2 mL of 1% lidocaine OR 1 mL of 4 mg/mL dexamethasone, 1 mL of 2% lidocaine and 1 mL saline injected into the plantar fascia
  Other Names: Cortisone
  Arms: Corticosteroid

SUMMARY:
This single-blinded, randomized-controlled trial compares the efficacy of ultrasound-guided onabotulinumtoxinA (BTX-A) injections to the flexor digitorum brevis with current standard of care corticosteroid injections to the plantar fascia for the treatment of refractory plantar fasciitis in patients that have failed six weeks of non-operative treatment.

DETAILED DESCRIPTION:
Treatment of plantar fasciitis is not well described in the current literature, often making management difficult for both providers and patients. Recent literature has suggested potential use of Onabotulinumtoxin A (BTX-A) as an effective treatment to reduce pain and allow patients to return to their previous level of functional activity. The study will consist of veteran patients at the George E Wahlen Department of Veteran's Affairs (SLC VA) in Salt Lake City, UT. This pilot study aims to randomize patients with plantar fasciitis into current standard of care treatment with corticosteroid injection into the plantar fascia and experimental treatment with BTX-A injection into the flexor digitorum brevis cohorts. We predict that those who receive BTX-A injections will report better outcomes on the Numeric Pain Rating Scale (NPRS) as well as the Foot and Ankle Ability Measure (FAAM) when compared to those receiving corticosteroid. The results of this study could aid in providing evidence towards more reliable and beneficial treatment of plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed increased pain when pressure applied at the medial calcaneal tubercle
2. X-ray negative for calcaneal fractures or tumors
3. Patient with plantar fasciitis who have failed 6 weeks of non-operative treatment

Exclusion Criteria:

1. Prior botulinum toxin injections in the plantar fascia
2. Any botulinum toxin injections in the past 3 months
3. Cortisone injection in the plantar fascia in the previous 3 months
4. Previous surgery on the plantar fascia
5. Active workers compensation claim for plantar fasciitis
6. Active infection or fever
7. Botox or steroid allergy
8. Pregnancy
9. Current other treatment specific to the plantar fascia or intent to undergo during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Change in general pain levels | Baseline to 1 (primary endpoint), 3, and 6 months
  Measured via patient-reported Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Change in foot and ankle-induced difficulties with activities of daily living | Baseline to 1 (primary endpoint), 3, and 6 months
  Measured via patient-reported Foot and Ankle Ability Measure (FAAM)
Number of subjects dropping out for repeat injection or surgical intervention | Baseline to 1 (primary endpoint), 3, and 6 months
  Measure how long therapeutic relief lasts

CONTACTS AND LOCATIONS:
Overall Officials: Mikol Anderson, DPM, Principal Investigator — VA Salt Lake City Health Care System
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Utah, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05367271/ICF_000.pdf